CLINICAL TRIAL: NCT04565678
Title: A Phase 1, Open-label, Randomized 4-period Crossover Study to Assess the Relative Bioavailability and Effect of Food on the Coated Granule Formulation of Mitapivat in Healthy Subjects
Brief Title: A Study to Assess the Relative Bioavailability and Effect of Food on the Coated Granule Formulation of Mitapivat in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-019
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Sequence 1: ABCD (Experimental): Participants will receive Treatment A (mitapivat tablet, orally, under fasted conditions once on Day 1 of Period 1) followed by Treatment B (mitapivat coated granules, orally, under fasted conditions once on Day 1 of Period 2) followed by Treatment C (mitapivat coated granules, with a strawberry yogurt, orally once on Day 1 of Period 3) followed by Treatment D (mitapivat coated granules, with a chocolate pudding, orally once on Day 1 of Period 4). Each Treatment Period will be separated by a Washout Period of 7 days.
  Interventions: Drug: Mitapivat tablets; Drug: Mitapivat coated granules
- Treatment Sequence 2: BDAC (Experimental): Participants will receive Treatment B (mitapivat coated granules, orally, under fasted conditions once on Day 1 of Period 1) followed by Treatment D (mitapivat coated granules, with a chocolate pudding, orally once on Day 1 of Period 2) followed by Treatment A (mitapivat tablet, orally, under fasted conditions once on Day 1 of Period 3) followed by Treatment C (mitapivat coated granules, with a strawberry yogurt, orally once on Day 1 of Period 4). Each Treatment Period will be separated by a Washout Period of 7 days.
  Interventions: Drug: Mitapivat tablets; Drug: Mitapivat coated granules
- Treatment Sequence 3: CADB (Experimental): Participants will receive Treatment C (mitapivat coated granules, with a strawberry yogurt, orally once on Day 1 of Period 1) followed by Treatment A (mitapivat tablet, orally, under fasted conditions once on Day 1 of Period 2) followed by Treatment D (mitapivat coated granules, with a chocolate pudding, orally once on Day 1 of Period 3) followed by Treatment B (mitapivat coated granules, orally, under fasted conditions once on Day 1 of Period 4). Each Treatment Period will be separated by a Washout Period of 7 days.
  Interventions: Drug: Mitapivat tablets; Drug: Mitapivat coated granules
- Treatment Sequence 4: DCBA (Experimental): Participants will receive Treatment D (mitapivat coated granules, with a chocolate pudding, orally once on Day 1 of Period 1) followed by Treatment C (mitapivat coated granules, with a strawberry yogurt, orally once on Day 1 of Period 2) followed by Treatment B (mitapivat coated granules, orally, under fasted conditions once on Day 1 of Period 3) followed by Treatment A (mitapivat tablet, orally, under fasted conditions once on Day 1 of Period 4). Each Treatment Period will be separated by a Washout Period of 7 days.
  Interventions: Drug: Mitapivat tablets; Drug: Mitapivat coated granules

INTERVENTIONS:
Drug: Mitapivat tablets — Oral tablets
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate
Drug: Mitapivat coated granules — Oral coated granules
  Other Names: AG-348; AG-348 sulfate hydrate; Mitapivat sulfate

SUMMARY:
The primary purpose of this study is to assess the relative bioavailability of the mitapivat coated granule formulation compared to the tablet formulation following a single oral dose of mitapivat under fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kilograms per square meter (kg/m^2), inclusive;
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations;
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception;
* Participant has no clinically significant history or presence of ECG findings as judged by the Investigator at Screening and Check-in.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator;
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, including the 2 soft foods administered in this study, or other substance, unless approved by the Investigator;
* History of stomach or intestinal surgery or resection including cholecystectomy that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed);
* History of any malignancy with the exception of non-melanomatous skin cancer in situ, cervical carcinoma in situ, or breast carcinoma in situ;
* Participant has liver function tests including alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, and total bilirubin that are greater than the upper limit of normal at Screening or Check-in;
* Participant has platelet count or hemoglobin and hematocrit values that are below the lower limit of normal at Screening or Check-in;
* Confirmed (eg, original value and 2 consecutive repeat measurements) systolic blood pressure >150 or <90 millimeters of mercury (mmHg), diastolic blood pressure >90 or <50 mmHg, and pulse rate >100 or <45 beats per minute (bpm);
* Confirmed QT interval corrected for heart rate using Fridericia's method (QTcF) >450 milliseconds (msec) (male participants) or >470 msec (female participants);
* History of active alcoholism or drug/chemical abuse within 2 years prior to Check-in;
* Alcohol consumption of >21 units per week for males and >14 units for females;
* Positive urine drug screen at Screening or positive alcohol breath test result or positive urine drug screen at Check-in;
* Positive hepatitis panel and/or positive human immunodeficiency virus test;
* Participants with an active infection requiring systemic antimicrobial therapy, or with an active infection deemed clinically significant by the Investigator during Screening;
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to dosing (whichever is longer);
* Participant has used any over-the-counter medications, including herbal or nutritional supplements, within 28 days (or 5 half-lives, whichever is longer) before the first dose of study drug until after the Follow up phone call;
* Participant has used any prescription (excluding hormone replacement therapy and hormonal birth control) medications within 30 days (or 5 half-lives, whichever is longer) before the first dose of study drug until after the Follow up phone call;
* Use of tobacco- or nicotine-containing products including cigarettes, snuff, nicotine patch, nicotine chewing gum, vaporizers, or inhalers, within 6 months prior to Screening until after the Follow up phone call, or positive cotinine at Screening or Check-in;
* Participant must refrain from marijuana or cannabinol-containing products for 7 days before Screening until after the Follow up phone call;
* Ingestion of poppy seed within 7 days prior to Check-in until after the Follow up phone call;
* Participant has consumed grapefruit or grapefruit juice, Seville orange, or Seville orange containing products (eg, marmalade) within 7 days before the first dose of study drug until after the Follow up phone call;
* Participant has consumed caffeine- or xanthine-containing products within 24 hours prior to first dose of study drug until after the Follow up phone call;
* Participant has consumed vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, and mustard), or charbroiled meats for 7 days prior to first dose of study drug until after the Follow-up phone call;
* Participant is involved in strenuous activity or contact sports from 7 days before Check-in until after the Follow-up phone call;
* Receipt of blood products within 2 months prior to Check-in;
* Participant has donated blood or blood products >450 milliliters (mL) within 30 days before the first dose of study drug;
* Participant has a poor peripheral venous access;
* Have previously completed or withdrawn from this study or any other study investigating mitapivat sulfate, and have previously received the mitapivat sulfate;
* Participant has a history of allergy to sulfonamides (eg, co-trimoxazole antibiotic, silver sulfadiazine topical antibiotic for burn wounds) that has been characterized by acute hemolytic anemia, drug-induced liver injury, anaphylaxis, rash of erythema multiforme type, or Stevens-Johnson syndrome.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Mitapivat Under Fasted Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Quantifiable Concentration (AUC0-t) of Mitapivat Under Fasted Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-∞) of Mitapivat Under Fasted Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Time to Reach Maximum Observed Concentration (Tmax) of Mitapivat Under Fasted Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)

SECONDARY OUTCOMES:
Cmax of Mitapivat Under Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
AUC0-t of Mitapivat Under Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
AUC0-∞ of Mitapivat Under Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Tmax of Mitapivat Under Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Relative Bioavailability (Frel) Under Fasted and Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Area Under the Plasma Concentration-Time Curve from Time Zero to Twelve Hours (AUC0-12) of Mitapivat Under Fasted and Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Apparent Plasma Terminal Elimination Half-life (t½) of Mitapivat Under Fasted and Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Apparent Total Plasma Clearance (CL/F) of Mitapivat Under Fasted and Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Apparent Volume of Distribution (Vz/F) of Mitapivat Under Fasted and Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Apparent Terminal Elimination Rate Constant (λz) of Mitapivat Under Fasted and Fed Conditions | Pre-dose and multiple time points post-dose (up to 72 hours)
Number of Participants With Adverse Event (AEs) | Up to approximately 9 weeks
Number of Participants With AEs, Graded by Severity | Up to approximately 9 weeks
Number of Participants With Clinically Significant Abnormal Clinical Laboratory Values | Up to approximately 9 weeks
Number of Participants With Clinically Significant Abnormal Findings for 12-lead Electrocardiogram (ECG) Parameters | Up to approximately 9 weeks
Number of Participants With Clinically Significant Abnormal Findings for Vital Signs Parameters | Up to approximately 9 weeks
Number of Participants With Clinically Significant Abnormal Physical Examination Findings | Up to approximately 9 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No